CLINICAL TRIAL: NCT01990118
Title: A Randomized, Multi-center, Open Label Trial to Establish the Therapeutic Equivalence Between Neoral® and Gengraf® in Stable Renal Allograft Recipients [Gengraf Conversion Study]
Brief Title: Gengraf Conversion Study in Stable Renal Allograft Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Ong Loke Meng, Consultant Nephrologist, Penang Hospital, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.041
Record Dates: First submitted 2010-03-04; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: End Stage Renal Failure
Keywords: Renal transplant; Renal allograft rejection; Cyclosporine; Gengraf
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoral (Active Comparator): Patients who continued to be treated with the drug Neoral.
  Interventions: Drug: Neoral
- Gengraf arm (Experimental): Patients were randomly selected to be converted to 'Gengraf® capsule containing 25mg or 100mg cyclosporine'
  Interventions: Drug: Gengraf® capsule containing 25mg or 100mg cyclosporine

INTERVENTIONS:
Drug: Neoral — Neoral® capsule containing 25mg or 100mg cyclosporine
  Other Names: Cyclosporine
  Arms: Neoral
Drug: Gengraf® capsule containing 25mg or 100mg cyclosporine — Transplant patients who were stable on Neoral were converted to Gengraf
  Other Names: Generic Cyclosporine
  Arms: Gengraf arm

SUMMARY:
The purpose of this study is to establish the therapeutic equivalence of Gengraf® with the standard treatment Neoral® for a treatment period of 6 months in stable renal allograft transplant recipients with respect to drug levels, dosage, and acute graft rejection and other adverse events.

DETAILED DESCRIPTION:
The introduction of cyclosporine (CsA) into clinical practice resulted in improvements in acute renal allograft rejection rate and graft survival in renal transplant patients. Gengraf a microemulsion formulation of CsA though granted an AB-rated equivalent to Neoral, because of concerns over the use of generic drugs in transplantation, we undertook this study to evaluate the clinical efficacy and safety of Gengraf.

We conducted a multicenter, randomized, open labeled study to establish the equivalence between Gengraf and Neoral in stable renal transplant recipients for a treatment period of 6 months. 6 months post transplant patients with stable graft function and receiving a stable dose of neoral were recruited into the study. Eligible patients were randomly assigned to remain on Neoral or convert to an equal milligram-for-milligram dose of Gengraf. The primary end-point was serum creatinine at 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from patient or parents/guardian.
2. Patients who are more than 6 months post transplant
3. Stable graft function i.e. serum creatinine less than 300 umol/l
4. Patients currently on a stable dose of capsule Neoral within last one month

Exclusion Criteria:

1. Multiple organ transplantation
2. Pregnant or nursing woman, or women of childbearing potential without an effective method of birth control. Effective birth control methods are oral contraception, Norplant, surgical sterilization, Intra Uterine Device or diaphragms in conjunction with spermicidal foam and condom on the male partner.
3. Participation in any drug trial in which the patient received an investigational drug within 30 days preceding the screening phase of this study.
4. Those persons directly involved in the conduct of the study.
5. Active infection at the time of screening for enrollment into trial.
6. Acute graft rejection within the past 3 months
7. Mentally unstable or history of mental diseases
8. History of drug or alcohol abuse within the past 2 years.
9. History of non-compliance to medical regimen and patients who are unwilling or unable to comply with the protocol.
10. Decompensated liver disease
11. Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2004-11; Primary Completion 2005-12 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Serum creatinine level at 12 weeks | at 12 weeks
  Serum creatinine level at 12 weeks after conversion from Neoral to Gengraf

SECONDARY OUTCOMES:
CsA trough concentration and at 2 hour after CsA administration, at 2 weeks, 6 weeks 12 weeks, 6 months, 9 months and 12 months post randomization. | weeks 2, 6, 12, months 6, 9 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Ong L Meng, MBBS, FRCP, Principal Investigator — Penang Hospital, Ministry of Health Malaysia
Locations (1):
- Clinical Research Centre, Penang Hospital, George Town, Pulau Pinang, Malaysia